CLINICAL TRIAL: NCT03292835
Title: Multicentric Non-Interventional Trial Evaluating Painless Hand Hygiene and LeiProtect® Dressing to Treat Complex Cutaneous Leishmaniasis in Algeria - LeiClean
Brief Title: Complex Cutaneous Leishmaniasis Healing Study in Algeria
Acronym: LeiClean
Status: Terminated | Type: Observational
Why Stopped: Production of LeiProtect suspended.
Sponsor: K. W. Stahl (Other)
Collaborators: Institut Pasteur (Industry); University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor-Investigator, K. W. Stahl, Prof. Dr. Dr., Waisenmedizin e. V. Promoting Access to Essential Medicine
Organization: Waisenmedizin e. V. Promoting Access to Essential Medicine (Other)
Other Study IDs: ALG 17/003
Record Dates: First submitted 2017-09-18; First posted 2017-09-26 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Cutaneous Leishmaniases
Keywords: complex; zoonotic; medical device
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Polymerase Chain Reaction (PCR). The differentiation of parasite species in between responders and eventual non-responders using sequencing technologies established in the Institute of Clinical Microbiology, Immunology and Hygiene, FAU Erlangen and University Hospital Erlangen.
  Smears with Giemsa staining.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: LeiProtect® — Filmogenic dressing gel
  Other Names: Alcohol Based Hand-Rub (ABHR)

SUMMARY:
This study evaluates the effect of clean wound management and dressing on complex zoonotic cutaneous leishmaniasis caused by L. major in the MENA region (Algeria). The patients will participate in the wound dressing themselves. The objective is to determine the amount of patients that can avoid systemic chemotherapy with pentavalent antimony which is compulsory for patients with complex CL lesions. In Algeria, this requires expensive hospital care because of the eventual toxic side effects of Sb(V).

DETAILED DESCRIPTION:
The investigator initiated, non-interventional LeiClean Trial with 100 CL patients presenting complex CL lesions, normally in need of a systemic an in-door treatment with meglumine antimoniate and in risk of systemic antimony toxicity (see inclusion criteria!) during the CL season of 2017/18 is part of the renewed cooperation treaty between the IPA and WM e. V. and originates from encouraging compassionate use observations after topical LeiClean treatment authorized by the Algerian Ministry of Health in December 2015. The study will be carried out in the ZCL region of M'Sila and Bou Saada.

The German Regulation Authority, BfArM, has granted a special approval according to §11 MPG (German regulation for Medical Devices) to the new filmogenic gel dressing LeiProtect®. The patients with complex cutaneous leishmaniasis (Giemsa and PCR confirmed) elected for indoor treatment with systemic antimony treatment are given the option for a LeiClean treatment of their lesions; they are instructed on hand hygiene and LeiProtect® dressing of their lesions which they carry out themselves at home during seven days. On day eight they come for lesion cleansing and photographic monitoring before they start another weekly LeiClean cycle. The patients can at any time opt for a conventional systemic chemotherapeutic treatment in a hospital if they are not satisfied with their healing progress. However, if the doctor realizes that after two months the hygienic wound management results in inadequate healing, he can also order hospital for the patients. The doctor will allow the patients to visualise their healing progress over the course of the trial through digital images on the computer.

After complete epithelisation of the lesions, the patients come for controls at monthly intervals up to a period of five months to check for eventual lesion relapses. The costs of the LeiClean outdoor treatment will be evaluated and compared to the already known hospital costs per patient for a three-week systemic indoor Sb(V) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject has Giemsa and PCR proven L.major cutaneous leishmaniasis
* Subject has complex zoonotic cutaneous leishmaniasis or Sb(V) incompatibility
* Subject gives voluntary consent

Exclusion Criteria:

* Immune deficiencies, skin tumours, allergy to 1,2-propylene glycol (rare)

Ages: 1 Week to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ZCL patients in the CL endemic region of M'Sila and Bou Saada, Algeria
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Lesion Epithelisation | 2 months
  Digital photo documentation

SECONDARY OUTCOMES:
No healing progress with LeiClean | 2 months
  Patients who have to be hospitalised for systemic Sb(V) treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zoubir Harrat, Dr., Principal Investigator — Pasteur Institute
Locations (1):
- NGO Waisenmedizin e. V., Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Organisation Homepage — http://www.waisenmedizin.org